CLINICAL TRIAL: NCT05532475
Title: Vitreous Level Of Tumor Necrosis Factor Alpha In Patients With Retinal Vein Occlusion
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Attya, Lecturer of ophthalmology- faculty of medicine- Cairo University, Kasr El Aini Hospital
Other Study IDs: MS-654-2021
Record Dates: First submitted 2022-09-03; First posted 2022-09-08 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Retinal Vein Occlusion
Keywords: Tumor necrosis factor alpha
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: patient with retinal vein occlusion
  Interventions: Diagnostic Test: measurement of vitreous level of tumor necrosis factor alpha
- control: cataract patient undergoing cataract surgery
  Interventions: Diagnostic Test: measurement of vitreous level of tumor necrosis factor alpha

INTERVENTIONS:
Diagnostic Test: measurement of vitreous level of tumor necrosis factor alpha — measurement of vitreous level of tumor necrosis factor alpha using ELISA technique

SUMMARY:
To assess the levels of TNF- α in vitreous samples of patients with retinal vein occlusion prior to administration of intravitreal anti-VEGF and compare them to levels in vitreous samples of normal subjects so as to investigate the association of vitreous tumor necrosis factor with the pathogenesis of retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with retinal vein occlusion not older than 6 months with no history of Anti-VEGF injection

Exclusion Criteria:

1. Diabetic patients.
2. Other causes of retinal vascular diseases.
3. Patients with history of treatment of retinal vein occlusion.
4. Previous intraocular surgery except cataract surgery performed 6 months before the study.
5. Subjects with severe systemic inflammatory diseases
6. Retinal vein occlusion secondary to retinal vasculitis.
7. All retinal pathologies.
8. Patients receiving Systemic steroids or Immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retinal venous occlusion patients admitted in KasrAlainy Hospital for Intravitreal Injection of Lucentis (Cases) compared to patient without retinal vein occlusion admitted for cataract surgery (Controls).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
to assess vitreous level of tumor necrosis factor alpha in retinal vein occlusion and compare it to patient undergoing cataract surgery | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr ALainy University hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No